CLINICAL TRIAL: NCT00188916
Title: A Clinical Comparison of Three Bronchial Blockers for One-Lung Ventilation in Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: UHN REB 04-0407-AE
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2006-09

CONDITIONS: Thoracic Surgery
Keywords: Bronchial blockers; Lung isolation; Thoracic Anesthesia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a clinical trial comparing surgical conditions during one-lung ventilation with three different bronchial blockers or with double-lumen endobronchial tubes.

ELIGIBILITY:
Inclusion Criteria:

* Left thoracotomy

Exclusion Criteria:

* Contraindication to lung isolation

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Slinger, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada